CLINICAL TRIAL: NCT02843724
Title: Integrative Care for Type 2 Diabetes: Evaluating the Impact of Naturopathic Adjunctive Care for Diabetic Patients of a Family Health Team
Brief Title: Integrative Care for Type 2 Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Responsible Party: Principal Investigator, Ellen Wong, Co Principal Investigator, The Canadian College of Naturopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanadianCNN
Record Dates: First submitted 2016-07-14; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Uncontrolled Type 2 Diabetes; HbA1c >7.0%
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Conventional) Arm (Active Comparator): Treatment of Type 2 Diabetes according to the Canadian Diabetes Association guidelines. Participants' other health concerns to be addressed as per usual care by practitioners at Wise-Elephant Family Health Team.
  Interventions: Other: Usual (Conventional) Care
- Integrative (Naturopathic + Conventional) Arm (Active Comparator): In addition to conventional care, participants will receive free naturopathic care at Brampton Naturopathic Teaching Clinic (located within the Brampton Civic Hospital). Senior student clinicians will provide care under the direct supervision of licensed naturopathic doctors. A naturopathic menu of treatment options have been designed to reflect naturopathic practice and vetted by 3 licensed naturopathic doctors and experts in the field. Participants' other health concerns will be addressed as per naturopathic doctors' discretion.
  Interventions: Other: Naturopathic Care; Other: Usual (Conventional) Care

INTERVENTIONS:
Other: Naturopathic Care — Naturopathic diabetes care will be selected from a pre-approved menu. Participants' other health concerns will be addressed at naturopathic doctors' discretion
  Arms: Integrative (Naturopathic + Conventional) Arm
Other: Usual (Conventional) Care — 2016 Canadian Diabetes Clinical Practice Guidelines (self-management, blood-glucose-lowering, vascular protection, pharmacotherapy) will be implemented

SUMMARY:
A two year, two arm pragmatic trial to investigate the integration of naturopathic care with conventional medical care to provide additional benefit beyond that of conventional medical care alone in achieving adequate control of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, enrolled as a patient with WE-FHT
* Ages 21-75 years old
* Diagnosed with type 2 diabetes and not adequately controlled (HbA1c > 7.0mmol/L)
* Currently seeking care with a medical doctor, nurse practitioner and/or physician assistant
* Willingness to adhere to randomized treatment with availability for follow-up
* Ability to answer self- and interviewer- administered questions in English or have an English speaking caregiver who can aid in answering self- and interviewer- administered questions
* Ability to provide written informed consent or give informed consent through substitute decision maker
* Capacity to maintain a diary and log of treatments and recommendations given during study

Exclusion Criteria:

* Lacking capacity for consent
* Pregnancy or an intention to become pregnant in the following two years
* Breastfeeding
* History of myocardial infarction within the past 6 months
* Chronic kidney (eGFR <30 mL/min) or liver disease
* Actively receiving care from a complex care diabetes clinic
* History of severe hypoglycemia in the last year resulting in hospital emergency care [where hypoglycemia is defined to be: 1) development of autonomic or neuroglycopenic symptoms, 2) low plasma glucose level (<4.0mmol/L for patients treated with insulin or an insulin secretagogue) and 3) symptoms responding to the administration of carbohydrate] or hypoglycemia unawareness
* Current bolus or pre-mixed insulin treatment
* Limited life expectancy (< 6 months)
* High level of functional dependency (inability to perform common activities of daily living)
* In participants aged 65yoa to 75yoa, the following also serve as exclusion criteria:

  1. Recent MI or stroke (within last 6 months)
  2. NYHA CHF Functional Capacity Stage III or above
  3. NYHA CHF Objective Assessment Stage C or greater (http://www.heart.org/HEARTORG/Conditions/HeartFailure/AboutHeartFailure/Classes-of-Heart-Failure_UCM_306328_Article.jsp)
  4. Planned revascularization procedure (PCI or coronary artery bypass graft) or coronary angiogram within 90 days after screening or randomization

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Clinically meaningful reduction of HbA1c above and beyond that of control arm | 1 year
  To assess the integration of naturopathic care to conventional medical care in obtaining a clinically meaningful reduction of HbA1c (equal or > 0.5%) above and beyond reduction of HbA1c in the control group of phase 1 at 52 week for participants from Wise Elephant Family Health Team (WE-FHT) with type 2 diabetes

SECONDARY OUTCOMES:
Incidence of metabolic syndrome | 2 year
Weight (as part of BMI) | 2 year
  Kg
Height (as part of BMI) | 2 year
  meters
Waist circumference (as part of metabolic syndrome) | 2 year
  inches
Fasting blood glucose | 2 year
  Fasting glucose (FG), biomarker associated with diabetes
Glycated hemoglobin (HbA1c) | 2 year
  Biomarker associated with diabetes
Blood pressure (BP) | 2 year
  Systolic and diastolic blood pressure, seated, resting
Total cholesterol (TC) (blood) | 2 year
  Biomarkers associated with cholesterol & cardiovascular risk
High-density lipoprotein (HDL-C) (blood) | 2 year
  Biomarkers associated with cholesterol & cardiovascular risk
Low-density lipoprotein (LDL-C) (blood) | 2 year
  Biomarkers associated with cholesterol & cardiovascular risk
Triglycerides (TG))(blood) | 2 year
  Biomarkers associated with cholesterol & cardiovascular risk
High-sensitivity C-reactive protein (hs-CRP) | 2 year
  Biomarker associated with cardiovascular risk
Incidence of smoking | 2 year
  Modifiable risk factors for cardiovascular disease
Incidence of obesity | 2 year
  Modifiable risk factors for cardiovascular disease, BMI equal to or greater than 30.0 kg/m2
Incidence of depression (PHQ-9) | 2 year
  Depression as defined by the PHQ-9
Impact on stress, anxiety, quality of life | 2 year
  ADDQol
Impact on anxiety | 2 year
  GAD 7
DES | 2 year
  Impact on quality of life
SF-12 | 2 year
  Impact on quality of life
Compliance/adherence with treatment prescriptions including changes in lifestyle, diet, exercise, and nutraceutical supplementation | 2 year
  Diet and physical activity tracker
Compliance/adherence with pharmaceutical prescriptions using a medication adherence questionnaire | 2 year
  MMAQ
Adverse Events | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Wong, ND, Principal Investigator — The Canadian College of Naturopathic Medicine
Locations (2):
- Canada (2):
  - Wise Elephant Family Health Team, Brampton, Ontario
  - The Canadian College of Naturopathic Medicine, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No